CLINICAL TRIAL: NCT02684838
Title: Vigilant ObservatIon of GlIadeL WAfer ImplaNT (VIGILANT) Registry: A Multicenter, Observational Registry to Collect Information on the Safety and Effectiveness of Gliadel® Wafer (Carmustine Implant) Used in Usual Medical Practice
Brief Title: Vigilant ObservatIon of GlIadeL WAfer ImplaNT Registry
Acronym: VIGILANT
Status: Completed | Type: Observational
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AR22.001
Record Dates: First submitted 2016-02-10; First posted 2016-02-18 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: CNS Tumor
Keywords: Gliadel, Carmustine wafer implant
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Available biomarker data will be collected (e.g., MGMT, EGFR, and IDH 1&2) and exploratory patient survival analysis will be conducted based upon biomarker status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational registry in patients who have been prescribed Gliadel Wafer by the physician as part of usual care.

DETAILED DESCRIPTION:
This is a prospective, observational registry in patients who have been prescribed Gliadel Wafer by the physician as part of usual care. Data will be collected on the safety and effectiveness of treatment with Gliadel Wafer perioperatively and ongoing during regular office visits up to 3-years. Patients enrolled in this registry will be asked to complete a questionnaire (Functional Assessment of Cancer Therapy-Brain [FACT-Br]) about their well-being and clinicians will complete the Karnofsky Performance Status (KPS) during office visits.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, by the patient or a legally acceptable representative, obtained before any registry-related activities are undertaken. The informed consent must be signed within 14 calendar days after surgery.
2. Male and female patients, greater than or equal to 18 years of age or age of majority in state of residence.
3. Patients planning to receive Gliadel Wafer, or having already received Gliadel Wafer and having signed consent to enroll in the registry within 14 calendar days after surgery for treatment of central nervous system (CNS) tumor(s), or are currently enrolled in another study where they received Gliadel Wafer.
4. Signed release form, by the patient or a legally acceptable representative, permitting abstraction of the patient's medical records at Baseline and during participation in the registry.

Exclusion Criteria:

1. The patient is enrolled in an interventional clinical trial, in which treatment for CNS tumor(s) is managed through a protocol that excludes Gliadel Wafer treatment.
2. Any abnormality or medical condition that, at the discretion of the Investigator, may put the patient at increased risk by participating in this registry.
3. Any other reason that, in the Investigator's opinion, makes the patient unsuitable to participate in this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been prescribed Gliadel Wafer by the physician as part of usual care
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall survival rate for patients treated with Gliadel Wafer | up to 3 years
  Time from Gliadel placement to death
To evaluate the disease-specific survival rate for patients treated with Gliadel Wafer | up to 3 years
  Time from Gliadel placement to death due to CNS tumor
To evaluate the progression-free survival rate for patients treated with Gliadel Wafer | up to 3 years
  Time from Gliadel placement to diagnosis of recurrent CNS tumor

SECONDARY OUTCOMES:
To evaluate the serious adverse events (SAEs) in patients treated with Gliadel Wafer. | up to 3 years
  Frequency of SAEs
To evaluate events of interest (EOI) in patients treated with Gliadel Wafer. | up to 3 years
  Frequency of EOIs
To evaluate nonserious, suspected adverse drug reactions (ADRs) in patients treated with Gliadel Wafer. | up to 3 years
  frequency of ADRs
To evaluate change in patient health status over time via patient reported outcomes (PRO) | up to 3 years
  Change in FACT-Br score from baseline to end of study participation
To evaluate change in patient health status over time via a practitioner/proxy reported scale | up to 3 years
  Change in KPS score from baseline to end of study participation
To evaluate the the reasons a physician does not insert Gliadel Wafers, in patients who were considered and consented for this Registry prior to the tumor resection procedure | up to 3 years
  reasons for screen failure

OTHER OUTCOMES:
To evaluate health care utilization though length of hospital stays for the primary procedure and any subsequent hospitalizations in patients treated with Gliadel Wafer | up to 3 years
  number of days in hospital following Gliadel insertion
To explore patient survival status based upon biomarker status. | up to 3 years

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Spine and Neuro Center, Huntsville, Alabama
  - Borrow Neurological Institute, Phoenix, Arizona
  - Spine Group Arizona At Honorhealth Scottsdale Osborn Medical Center, Scottdale, Arizona
  - Neurological Associates of Tucson, DBA Center for Neurosciences, Tucson, Arizona
  - David Geffen School of Medicine at UCLA; Departments of Neurosurgery and Pathology at the, Los Angeles, California
  - University of California, San Francisco Department of Neurological Surgery, San Francisco, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Baycare Medical Group, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Beacon Medical Group, Elkhart, Indiana
  - Baptist Health Paducah, Paducah, Kentucky
  - Oschner Medical Center, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - McLaren Bay Neurology Associates, Bay City, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Depaul Hospital, Bridgeton, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Western Regional Ctr for Brain and Spine Surgery, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Jfk Medical Center, Edison, New Jersey
  - Albany Medical Center Hospital, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Brain Tumor Center, Lake Success, New York
  - Crouse Neuroscience Institute, Syracuse, New York
  - Vidant Medical Center, Greenville, North Carolina
  - Wake Forest Baptist Med Center, Winston-Salem, North Carolina
  - Mount Carmel Neurosurgery, Columbus, Ohio
  - University of Oklahoma - Stevenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Grand Strand Medical Center, Myrtle Beach, South Carolina
  - University of Washington School of Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lillehei KO, Kalkanis SN, Liau LM, Mydland DE, Olson J, Paleologos NA, Ryken T, Johnson T, Scullin E. Rationale and design of the 500-patient, 3-year, and prospective Vigilant ObservatIon of GlIadeL WAfer ImplaNT registry. CNS Oncol. 2018 Apr;7(2):CNS08. doi: 10.2217/cns-2017-0036. Epub 2017 Dec 5. PMID 29206049